CLINICAL TRIAL: NCT00771277
Title: Team Based Initiative Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 08-383
Record Dates: First submitted 2008-10-08; First posted 2008-10-13 (Estimated); Results first posted 2014-09-18 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-08

CONDITIONS: Traumatic Brain Injury
Keywords: Brain Injuries; Caregivers; Volunteer Workers; Social Networks
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Use of volunteer support teams to provide services
  Interventions: Behavioral: Support Teams

INTERVENTIONS:
Behavioral: Support Teams — Use of volunteers organized into teams with a coordinator to provide services to TBI family

SUMMARY:
Traumatic brain injury (TBI) has been called the signature injury of the Iraq War. This pilot study investigated family needs of 6 rural families caring for a Veteran with TBI. Two Veterans had moderate TBI and all had comorbid post traumatic stress disorder diagnoses. The veterans were 1 to 5 years post-injury. Families were reluctant to include others in helping the family because of privacy concerns, desire for independence, and negative employment repercussions if the extent of the TBI deficit became known in the community. Most were still employed, despite TBI deficits. Despite having previously received information, families still had substantial needs for information about the condition and its prognosis and sequelae (e.g., why things happen, unsafe/frightening behaviors, work, finances, communication changes) and the availability and types of services (e.g., who to contact, benefits, help needed)

DETAILED DESCRIPTION:
Background/Rationale: Traumatic brain injury (TBI) has been called the signature injury of the Iraq War. This pilot study was an investigation of the feasibility of volunteer support teams for families providing care to a returning Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) veteran with TBI. Volunteer support teams coordinate tasks and effort for family and volunteers. This support model is particularly relevant for families in rural areas that are likely to be under-funded in home and community services.

Objectives: The original study objective was to determine feasibility of, and barriers to, implementing volunteer support teams with rural families of OEF/OIF veterans with recently diagnosed moderate-severe TBI. A secondary objective was to provide information on TBI to families and volunteers.

Methodology: The project coach met the family in the home to identify unmet needs and to determine availability of family and friends who could help meet needs. The coach provided training about TBI and a Resource Book with information on TBI diagnosis, prognosis, and symptoms. There were baseline, monthly, and study end qualitative interviews with the family focusing on concerns.

Findings/Result: Fifteen families were referred; TBI levels were mainly mild. Six families were enrolled. Two Veterans had moderate TBI and all had comorbid post traumatic stress disorder diagnoses. All lived in rural communities. The veterans were 1 to 5 years post-injury and support systems were already in place, although these systems were small. Families did not want to implement caregiving teams because of privacy concerns, desire for independence, and negative employment repercussions if the extent of the TBI deficit became known in the community. Most were still employed, despite TBI deficits. However, the project identified that families had substantial needs for information about the condition and its prognosis and sequelae (e.g., why things happen, unsafe/frightening behaviors, work, finances, communication changes) and the availability and types of services (e.g., who to contact, benefits, help needed). Families often reported feeling lost in negotiating the DoD and VA systems.

Impact: Issues and concerns for rural, mild TBI veterans and their families were identified. Families and the Veteran may not be ready to accept the diagnosis when it first occurs. Families and the veteran identified a need for just-in-time information on TBI, its consequences, and services available. The delicate balance between return to full functioning as a community member and the deficits of TBI is threatened by family independence, privacy needs, and fear of loss of employment. The study identified opportunities for community education and for coordination between the military and VHA.

ELIGIBILITY:
Inclusion Criteria:

* The primary family member caregiver of the Traumatic Brain Injury (TBI) veteran
* Veteran receiving care at the Memphis Veterans Affairs Medical Center
* Perceived need of help and support
* Willing to participate in the study after discussion with OEF/OIF Program
* Manager or team member

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Olivia Nichols, PhD, Principal Investigator — Memphis VA Medical Center, Memphis, TN
Locations (1):
- Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All families were National Guard families. The veterans were divided between mild and moderate TBI with co-morbid PTSD and 1 to 5 years post-injury. Patients were all male except for one wife. All were Caucasian. Ages of patients ranged from mid 20s to mid 40s.
Groups:
- Arm 1: Family experience of concerns and providing support to TBI patient
Arm/Group | Arm 1
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [32 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Relationship to patients [Number; unit: participants]
  wife | 4
  husband | 1
  grandmother | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported 5 Themes
Description: Six caregivers of TBI patients were interviewed; responses were transcribed and coded; inter-rater agreement was calculated. Themes were lack of understanding about TBI and its long-term effects and the differences between TBI and PTSD, privacy concerns, independence, fear of negative employment/financial repercussions, and difficulty in interactions with the Department of Defense (DoD) and the Department of Veterans Affairs (VA)
Time Frame: collected over 3 interviews of approximately 1 hour each
Measure: Number; unit: participants
Groups:
- TBI Caregivers: Family caregivers providing support to TBI patients.
Arm/Group | TBI Caregivers
Number analyzed (Participants) | 6
participants
  Lack of information and need for information | 6
  Privacy concerns | 6
  Independence of family | 6
  fear of negative employment/financial repercussion | 6
  difficulty in interactions with DoD and VA | 6

2. Secondary Outcome: PHQ-9
Description: The Patient Health Questionnaire (PHQ-9) (Kroenke, Spitzer, & Williams, 2001) assesses caregiver depression and anxiety on a scale from not at all (0) to nearly every day (3), with higher total scores indicating greater symptoms. Scores range from 0-27. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression respectively.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TBI Caregivers
Number analyzed (Participants) | 6
units on a scale | 11.5 (6.8)

3. Secondary Outcome: Zarit Burden Inventory
Description: Caregiver burden, as measured by the 12-item Zarit Burden Interview (Bédard et al., 2001; Zarit, Reever, & Bach-Peterson J, 1980). Burden includes concepts such as lack of time because of care, strain, restriction of life, etc. Items are scored from never (0) to nearly always (4), and higher total scores indicate greater burden. Total scores range from 0 to 88.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TBI Caregivers
Number analyzed (Participants) | 6
units on a scale | 23.0 (6.7)

ADVERSE EVENTS:
Description: Adverse Events were not collected/assessed in this study.
Arm/Group | TBI Caregivers
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No